CLINICAL TRIAL: NCT04070508
Title: Early Detection of Advanced Liver Fibrosis in Patients With Excessive Alcohol Intake
Brief Title: Early Detection of Alcoholic Liver Disease
Status: Withdrawn | Type: Observational
Why Stopped: Staff in the lab have transitioned to a new institution so there are no personnel available to recruit or resume the study.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ramon Bataller, Principal Investigator, University of Pittsburgh
Other Study IDs: STUDY19020346
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Alcoholic Liver Disease; Alcoholic Fibrosis of Liver; Alcoholic Cirrhosis; Excessive Drinking; Alcohol Abuse; Alcohol Use Disorder; Alcohol Dependence; Alcohol-Related Disorders
Keywords: early detection; alcoholic liver disease; alcohol
MeSH Terms: conditions — Liver Diseases, Alcoholic; Liver Cirrhosis, Alcoholic; Alcoholism; Alcohol-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — The samples collected in this study including blood, urine, liver tissue and saliva.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study to identify the prevalence of advanced liver fibrosis among patients with excessive alcohol intake using a non-invasive method (FibroScan®) and to characterize the main environmental, genetic and epigenetic factors that could influence the development of advanced fibrosis.

The investigators will include patients 21 years of age or older with excessive alcohol intake, with abnormal AST, ALT, GGT and/or bilirubin, and without any evidence of decompensated liver disease (jaundice, ascites, encephalopathy).

Liver fibrosis will be estimated by FibroScan®. A designed questionnaire for studying environmental and psychosocial factors will be filled by the included patients, and blood samples will be obtained to study genetic and epigenetic factors.

The patients with advance fibrosis will be referred to the specialist for surveillance and treatment according to current clinical guidelines.

DETAILED DESCRIPTION:
Background:

The Global Status Report on Alcohol and Health 2014 from the World Health Organization indicates that alcohol abuse accounts for 50% of cirrhosis worldwide. Therefore, alcoholic liver disease (ALD) is a main cause of advanced liver fibrosis globally. ALD encompasses a range of disorders including simple steatosis, alcoholic steatohepatitis, fibrosis, cirrhosis, and hepatocellular carcinoma. In addition, patients with underlying ALD and active drinking can develop an episode of acute-on-chronic liver injury called "alcoholic hepatitis", which portends a poor prognosis.

Most patients with ALD are identified during the late stages of the disease when liver decompensation occurs. In fact, a recent global epidemiologic study (GLADIS) showed that ALD is by far the liver disease that is detected at the latest stages (ratio of early/late referral negative 8-fold). These results strongly suggest that there is a dire need for the early detection of ALD patients, which currently is almost nonexistent.

A non-invasive method to screen for advanced fibrosis and cirrhosis is transient elastography (FibroScan®). This modality could potentially diagnose silent liver disease among heavy drinkers, allowing for earlier referral to a specialty liver clinic for further treatment.

Individual susceptibility to the development of advanced fibrosis among heavy drinkers is likely determined by a combination of environmental, genetic and epigenetic factors, yet the mechanisms are largely unknown.

Exposing the exact risk factors for the progression of subclinical liver disease to advanced fibrosis and cirrhosis among heavy alcohol users may assist with prognostication and help influence a patient's decision to abstain from alcohol.

The main goal of this study is to identify the prevalence of advanced liver fibrosis (F3 y F4) among patients with excessive alcohol intake using a non-invasive method (FibroScan®) and refer those who already have evidence of advanced fibrosis (F3-4 stage) to a specialized ALD clinic for treatment. The secondary goal is, to identify the main psychosocial, environmental, genetic and epigenetic factors that influence the individual susceptibility to develop advanced ALD and design a risk algorithm taking into account the interaction between these factors.

Design: This is a prospective observational single center study.

Length of participation:

* Subjects without detection of advanced fibrosis: no follow-up requiered.
* Subjects with detection of advanced fibrosis: these patients will be referred to the specialist for surveillance. In this group of patients, the investigators will record the visits every six months as standard of care during the first year, and in each visit, a questionnaire will be performed.

End of the study: The duration of the project is expected to be two years.

Study development: Patients will be recruited within UPMC Presbyterian (Oakland) and UPMC McKeesport.

Study procedures:

- Screening procedure: Those patients willing to participate in the study will sign the informed consent before screening process. In this process, inclusion and exclusion criteria will be checked.

* Clinical and anthropometric data
* Questionnaire
* FibroScan®
* Blood, liver tissue, urine and saliva collection and testing

Statistics:

General features and characteristics of the analysis:

Descriptive statistics will be used to report baseline characteristics of our study population as well as the incidence and prevalence of variables of interest. Chi-square test will be used to compare frequency distributions between subgroups for categorical variables. Mann-Whitney U will be used to compare continuous variables when variables do not follow normal distributions. Univariate analyses, using Chi-square, Student's t-test and Mann-Whitney U test will be used to assess the association between potential factors and advanced fibrosis. Logistic regression models will be fitted to select the best subset of predictors for advanced fibrosis. Those factors showing a clinically and statistically significant association with the outcome in univariate analyses will be selected for the initial models. The final models will be fitted by using a step-wise forward method based on model Likelihood Ratios with the same significance level (p<0.05) for entering and dropping variables. The significance level will be set at p<0.05 for all the analyses. Statistical analyses will be performed using IBM SPSS Statistics.

Sample size:

The investigators calculated a sample size of 350 subjects. An interim analysis will be performed.

Direct access to data source:

Clinical data will be collected into a web-based and HIPAA-compatible database system. The information will be registered in the electronic record system, Research Electronic Data Capture (REDCap), which has been validated by the ERIS / EDC Support team to ensure HIPAA compliance. REDCap is also assessed by the Partners Information Security Risk Assessment Team to ensure compliance with all Partners HealthCare policies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with an alcohol use disorder (AUD) identification test (AUDIT) with a total score of 8 or more or patients with a score lower than 8 in the AUDIT test but for whom there is a high suspicion of current or recent (within one year) AUD based on medical history or self-reported history of excessive alcohol use, stigmata of alcohol use on physical exam, liver chemistry abnormalities, and/or alcohol-induced organ involvement other than decompensated liver disease.
* Patients who admit having a persistent alcohol intake of more than 40 g/daily for women and 60 g/daily for men.
* Patients with abnormal AST, ALT, GGT and/or bilirubin.
* 21 years of age or older.
* Signed informed consent.

Exclusion Criteria:

* Patients with a history of liver disease or decompensated advanced liver disease (i.e: jaundice episodes, ascites, hepatic encephalopathy, variceal bleeding, hepatorenal syndrome) or known hepatocellular carcinoma.
* Patients with severe extrahepatic disease or terminal illness.
* Patients who are pregnant or breast-feeding. However, pre-menopausal women capable of bearing children will be allowed to participate in the study provided they have a reliable method of birth control and have a negative pregnancy test prior to inclusion.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 21 years of age or older with excessive alcohol intake, with abnormal AST, ALT, GGT and/or bilirubin, and without any evidence of decompensated liver disease (jaundice, ascites, encephalopathy).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-10-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Advanced fibrosis and cirrhosis assessed by FibroScan | baseline
  Prevalence of advanced liver fibrosis and cirrhosis among patients with excessive alcohol intake using FibroScan.
  Cut-off value for advanced fibrosis (F3) >8 kPa.

CONTACTS AND LOCATIONS:
Overall Officials: RAMON BATALLER, MD, PhD, Principal Investigator — University of Pittsburgh

REFERENCES:
- [Background] Shah ND, Ventura-Cots M, Abraldes JG, Alboraie M, Alfadhli A, Argemi J, Badia-Aranda E, Arus-Soler E, Barritt AS 4th, Bessone F, Biryukova M, Carrilho FJ, Fernandez MC, Dorta Guiridi Z, El Kassas M, Eng-Kiong T, Queiroz Farias A, George J, Gui W, Thurairajah PH, Hsiang JC, Husic-Selimovic A, Isakov V, Karoney M, Kim W, Kluwe J, Kochhar R, Dhaka N, Costa PM, Nabeshima Pharm MA, Ono SK, Reis D, Rodil A, Domech CR, Saez-Royuela F, Scheurich C, Siow W, Sivac-Burina N, Dos Santos Traquino ES, Some F, Spreckic S, Tan S, Vorobioff J, Wandera A, Wu P, Yacoub M, Yang L, Yu Y, Zahiragic N, Zhang C, Cortez-Pinto H, Bataller R. Alcohol-Related Liver Disease Is Rarely Detected at Early Stages Compared With Liver Diseases of Other Etiologies Worldwide. Clin Gastroenterol Hepatol. 2019 Oct;17(11):2320-2329.e12. doi: 10.1016/j.cgh.2019.01.026. Epub 2019 Jan 29. PMID 30708110
- [Background] Altamirano J, Bataller R. Alcoholic liver disease: pathogenesis and new targets for therapy. Nat Rev Gastroenterol Hepatol. 2011 Aug 9;8(9):491-501. doi: 10.1038/nrgastro.2011.134. PMID 21826088
- [Background] Raynard B, Balian A, Fallik D, Capron F, Bedossa P, Chaput JC, Naveau S. Risk factors of fibrosis in alcohol-induced liver disease. Hepatology. 2002 Mar;35(3):635-8. doi: 10.1053/jhep.2002.31782. PMID 11870378
- [Background] Lackner C, Spindelboeck W, Haybaeck J, Douschan P, Rainer F, Terracciano L, Haas J, Berghold A, Bataller R, Stauber RE. Histological parameters and alcohol abstinence determine long-term prognosis in patients with alcoholic liver disease. J Hepatol. 2017 Mar;66(3):610-618. doi: 10.1016/j.jhep.2016.11.011. Epub 2016 Nov 25. PMID 27894795
- [Background] Muntaner L, Altamirano JT, Augustin S, Gonzalez A, Esteban R, Guardia J, Genesca J. High doses of beta-blockers and alcohol abstinence improve long-term rebleeding and mortality in cirrhotic patients after an acute variceal bleeding. Liver Int. 2010 Sep;30(8):1123-30. doi: 10.1111/j.1478-3231.2010.02287.x. Epub 2010 Jun 1. PMID 20536715
- [Background] Mueller S, Seitz HK, Rausch V. Non-invasive diagnosis of alcoholic liver disease. World J Gastroenterol. 2014 Oct 28;20(40):14626-41. doi: 10.3748/wjg.v20.i40.14626. PMID 25356026
- [Background] Buch S, Stickel F, Trepo E, Way M, Herrmann A, Nischalke HD, Brosch M, Rosendahl J, Berg T, Ridinger M, Rietschel M, McQuillin A, Frank J, Kiefer F, Schreiber S, Lieb W, Soyka M, Semmo N, Aigner E, Datz C, Schmelz R, Bruckner S, Zeissig S, Stephan AM, Wodarz N, Deviere J, Clumeck N, Sarrazin C, Lammert F, Gustot T, Deltenre P, Volzke H, Lerch MM, Mayerle J, Eyer F, Schafmayer C, Cichon S, Nothen MM, Nothnagel M, Ellinghaus D, Huse K, Franke A, Zopf S, Hellerbrand C, Moreno C, Franchimont D, Morgan MY, Hampe J. A genome-wide association study confirms PNPLA3 and identifies TM6SF2 and MBOAT7 as risk loci for alcohol-related cirrhosis. Nat Genet. 2015 Dec;47(12):1443-8. doi: 10.1038/ng.3417. Epub 2015 Oct 19. PMID 26482880
- [Background] Bataller R, Gao B. Liver fibrosis in alcoholic liver disease. Semin Liver Dis. 2015 May;35(2):146-56. doi: 10.1055/s-0035-1550054. Epub 2015 May 14. PMID 25974900
- [Background] Moran-Salvador E, Mann J. Epigenetics and Liver Fibrosis. Cell Mol Gastroenterol Hepatol. 2017 Apr 26;4(1):125-134. doi: 10.1016/j.jcmgh.2017.04.007. eCollection 2017 Jul. PMID 28593184
- [Background] Singal AK, Bataller R, Ahn J, Kamath PS, Shah VH. ACG Clinical Guideline: Alcoholic Liver Disease. Am J Gastroenterol. 2018 Feb;113(2):175-194. doi: 10.1038/ajg.2017.469. Epub 2018 Jan 16. PMID 29336434